CLINICAL TRIAL: NCT02224742
Title: LeucoPatch in the Management of Hard-to-heal Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12EN005; ISRCTN27665670 (Other: ISRCTN)
Record Dates: First submitted 2014-08-22; First posted 2014-08-25 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LeucoPatch (Experimental): Usual care supplemented by the application of LeucoPatch centrifugates that comprise autologous fibrin patches containing living white cells and platelets
  Interventions: Device: LeucoPatch
- Usual care (Active Comparator): Usual care provided in a multidisciplinary foot care clinic, in accordance with international guidelines
  Interventions: Other: Usual care

INTERVENTIONS:
Device: LeucoPatch — LeucoPatch® is prepared by centrifuging one or more 18mL aliquots of the participant's venous blood in the LeucoPatch device and bench-top centrifuge. The centrifugation yields a tough layer of fibrin, with viable white cells and platelets, and this is applied directly to the wound surface using sterile forceps. The wound is then covered with an inert primary dressing, secondary protective dressing and the ulcerated area protected with appropriate off-loading. The patch is prepared and applied each week for up to 20 weeks or until the wound is judged healed.
  Arms: LeucoPatch
Other: Usual care — Usual wound care provided in a multidisciplinary foot care clinic , in accordance with international guidelines.
  Components of usual wound care include:
  * Formal assessment of ulcer and surrounding skin
  * Provision of any necessary off-loading
  * Debridement (i) sharp, (ii) other as appropriate (but excluding the use of larvae)
  * Appropriate dressing products
  * Appropriate antibiotic therapy
  * Nutrition and self care
  * Optimal glycaemic control
  * Revascularisation if deemed clinically necessary
  * Continued close observation
  Arms: Usual care

SUMMARY:
Diabetic foot ulcers are the source of considerable suffering and cost and there are currently no wound care products available that have been demonstrated to improve healing, or that are cost effective. There have however been a small number of studies which have examined the use of platelets or fluid derived from platelets, either from the patient's own blood or from blood bank products. These have suggested some promise, but have suffered from technical difficulties in making a suitable wound care product or the volume of blood required to derive the product. It is thought that the reason why they may work is that growth factors released by the platelets may stimulate the wound to heal.

This study will be a formal, randomised controlled trial to assess a new device for creating a wound care product which is a plug or patch comprising fibrin, white cells and platelets derived from 18 mls of the patients own blood. The application of this fibrin/white cell/platelet patch to the patients wound on a weekly basis will be compared with usual best care in patients with hard to heal Diabetic Foot Ulcers in a secondary care setting in 25 centres in the United Kingdom, Denmark and Sweden.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 years and over who have diabetes complicated by one or more ulcers on a foot or both feet below the level of the malleoli, excluding ulcers confined to the interdigital cleft.
* Those with more than one eligible ulcer will have one - usually the largest or more clinically significant - selected at screening as the index ulcer.
* Eligible ulcers will be hard-to-heal, meaning that the cross-sectional area will decrease by less than 50 % during a four week run-in period.
* The cross-sectional area of the index ulcer will be ≥50 and ≤1000 mm2 at the end of the 4 week run-in period.
* At randomisation, the index ulcer will be clinically non-infected according to IDSA criteria
* Either the ankle-brachial index (ABPI) in the affected limb will be between 0.50 and 1.40 or the dorsalis pedis pulse and/or tibialis posterior pulse will be palpable.
* HbA1c ≤108 mmol/mol at screening
* Participants will have the capacity to understand study procedures, and will be able to provide written informed consent.

Exclusion Criteria:

* Haemoglobin concentration <105 g/L or 6.5 mmol/L at screening.
* Presence of sickle-cell anaemia, haemophilia, thrombocytopenia (<100x109/L) or other clinically significant blood dyscrasia
* Known potential infectivity of blood products, including known HIV and hepatitis
* Dialysis or an estimated GFR (based on cystatine C or serum creatinine) <20 ml/min/1.73m2
* Increase in cross-sectional area of the index ulcer by ≥25% during the 4 week run-in period, or is either smaller than 50 mm2 or larger than 1000 mm2 at the end of that time.
* Clinical signs of infection of the index ulcer or reason to suspect that infection is present at randomisation.
* Revascularisation procedure in the affected limb planned, or undertaken within the preceding 4 weeks.
* Current treatment with cytotoxic drugs or with systemically administered glucocorticoids or other immunosuppressants.
* Treatment of foot ulcers with growth factors, stem cells or equivalent preparation within the preceding 8 weeks
* The need for continued use of negative pressure wound therapy
* Likely inability to comply with the need for weekly visits because of planned activity.
* Participation in another interventional clinical foot ulcer-healing trial within last the 4 weeks at the time of screening.
* Prior randomisation in this trial.
* Judgement by the investigator that the patient does not have the capacity to understand the study procedures or provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Healing | Within 20 weeks of randomisation
  Healing will be defined as complete epithelialisation without discharge that is maintained for 4 weeks and is confirmed by an observer blind to randomisation group.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Game, FRCP, Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust
Locations (32):
- Denmark (7):
  - Steno Diabetes Center, Gentofte Municipality
  - Herlev Hospital, Herlev
  - Nordsjællands Hospital, Hillerød
  - Kolding Sygehus, Kolding
  - Bispebjerg Hospital, København NV
  - Odense University Hospital, Odense
  - Viborg Sårcenter, Viborg
- Sweden (3):
  - Centralsjukhuset Kristianstad, Kristianstad
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Solna
- United Kingdom (22):
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - South Devon Healthcare NHS Foundation Trust, Torquay, Devon
  - The Ipswich Hospital NHS Trust, Ipswich, Suffolk
  - The Mid Yorkshire Hospitals NHS Trust, Pontefract, West Yorkshire
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Lancashire Teaching Hospitals NHS Foundation Trust, Chorley
  - Dartford and Gravesham NHS Trust, Dartford
  - Derby Hospitals NHS Foundation Trust, Derby
  - The Dudley Group NHS Foundation Trust, Dudley
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Gateshead Health NHS Foundation Trust, Gateshead
  - Harrogate and District NHS Foundation Trust, Harrogate
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHSTrust, Leicester
  - United Lincolnshire Hospitals NHS Trust, Lincoln
  - Norwich and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Berkshire NHS Foundation Trust, Reading
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - City Hospitals Sunderland NHS Foundation Trust, Sunderland
  - Royal Wolverhampton Hospitals NHS Trust, Wolverhampton

REFERENCES:
- [Derived] Game F, Jeffcoate W, Tarnow L, Jacobsen JL, Whitham DJ, Harrison EF, Ellender SJ, Fitzsimmons D, Londahl M; LeucoPatch II trial team. LeucoPatch system for the management of hard-to-heal diabetic foot ulcers in the UK, Denmark, and Sweden: an observer-masked, randomised controlled trial. Lancet Diabetes Endocrinol. 2018 Nov;6(11):870-878. doi: 10.1016/S2213-8587(18)30240-7. Epub 2018 Sep 19. PMID 30243803